CLINICAL TRIAL: NCT06529224
Title: Social Egg Freezing: Will Health Professionals Offer it ?
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN942023/CHUSTE
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Infertility,Female
Keywords: Elective egg freezing; Attitude of health professionals; Health knowledge; Aging; Female infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health professionals: General practitioner, gynecologist or midwife
  Interventions: Other: Online questionnaire

INTERVENTIONS:
Other: Online questionnaire — An online questionnaire will be distributed in electronic format to all the healthcare professionals concerned.

SUMMARY:
In 2021, the revision of bioethics laws opened the door to elective egg freezing. This gives women, between their 29th and 37th birthdays, the opportunity to freeze their eggs in order to combat age decline fertility. However, communication about this new possibility has remained limited both toward women and their health professional.

DETAILED DESCRIPTION:
Thus, the hypothesize of this study is that these professionals, namely physicians, gynecologists and midwives, are insufficiently aware of age-related fertility decline and unaware of the possibility of elective egg freezing.

This multicenter observational cross-sectional study whose objective will be:

* To assess the knowledge of these professionals in terms of age-related fertility decline.
* To measure their propensity to spontaneously broach the subject with their childless patients.
* To assess their knowledge and support for elective egg freezing. This study will be done using an online questionnaire that will be distributed in electronic format to all the health professionals concerned in the participating areas.

This study will provide valuable knowledge on the perception of elective egg freezing by health professionals, determine their training needs and motivate new information campaigns on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Be a general practitioner, gynecologist or midwife in practice for at least one year
* Follow patients between 29 and 37 years old (for their contraception for example)

Exclusion Criteria:

* Have been practising for less than a year
* Have no patients aged between 29 and 37

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Practising GPs, gynaecologists or midwives
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Knowledge of primary care professionals regarding age-related decline in fertility. | Day 1
  Analysis questionnaire results.
Propensity to spontaneously broach the subject with their patients without children. | Day 1
  Analysis questionnaire results.
Knowledge and support for the elective egg freezing. | Day 1
  Analysis questionnaire results.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe KLEIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No